CLINICAL TRIAL: NCT01881711
Title: An Operator-Blinded Study of the Efficacy of ShuntCheck-Micro-Pumper, a Non-Invasive Diagnostic Procedure, in Detecting Ventricular Shunt Patency or Occlusion and in Predicting Clinical Outcome in Children and Adolescents Presenting to Emergency Departments and Neurosurgery Clinics
Brief Title: ShuntCheck-Micro-Pumper Pediatric Clinical Outcomes Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: NeuroDx Development (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: NDxDev-SCMP-2013; R44NS067772 (NIH)
Record Dates: First submitted 2013-06-13; First posted 2013-06-20 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Suspected CSF Shunt Obstruction
Keywords: hydrocephalus; CSF shunt; shunt malfunction; shunt obstruction; ShuntCheck; ShuntCheck-Micro-Pumper
MeSH Terms: conditions — Hydrocephalus | interventions — Diagnostic Imaging; Tomography, X-Ray Computed

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- SCMP plus Imaging (Experimental): SCMP plus Imaging will be compared to clinical outcomes within 7 days of ED/NC visit - either shunt obstruction confirmed during shunt revision surgery or shunt patency confirmed by no surgery or patency confirmed in surgery.
  Interventions: Device: ShuntCheck-Micro-Pumper (SCMP); Device: Imaging
- Imaging Alone (Active Comparator): Imaging alone will be compared to clinical outcomes within 7 days of ED/NC visit - either shunt obstruction confirmed during shunt revision surgery or shunt patency confirmed by no surgery or patency confirmed in surgery.
  Interventions: Device: Imaging
- SCMP Rule Out for Low Risk Cases (Experimental): SCMP results in patients judged by the physician to be "Unlikely to require shunt surgery" will be compared to clinical outcomes within 7 days of ED/NC visit - either shunt obstruction confirmed during shunt revision surgery or shunt patency confirmed by no surgery or patency confirmed in surgery - to determine Negative Predictive Value in ruling out shunt malfunction
  Interventions: Device: ShuntCheck-Micro-Pumper (SCMP)
- Imaging Rule for Low Risk Cases (Active Comparator): Imaging results in patients judged by the physician to be "Unlikely to require shunt surgery" will be compared to clinical outcomes within 7 days of ED/NC visit - either shunt obstruction confirmed during shunt revision surgery or shunt patency confirmed by no surgery or patency confirmed in surgery - to determine Negative Predictive Value in ruling out shunt malfunction
  Interventions: Device: Imaging
- SCMP plus Imaging in Uncertain Cases (Experimental): SCMP plus imaging results in patients who are admitted for observation results in patients judged by the physician to be "Unlikely to require shunt surgery" will be compared to clinical outcomes within 7 days of ED/NC visit - either shunt obstruction confirmed during shunt revision surgery or shunt patency confirmed by no surgery or patency confirmed in surgery - to determine Positive and Negative Predictive Value
  Interventions: Device: ShuntCheck-Micro-Pumper (SCMP); Device: Imaging
- Imaging alone in Uncertain Cases (Active Comparator): Imaging results in patients who are admitted for observation results in patients judged by the physician to be "Unlikely to require shunt surgery" will be compared to clinical outcomes within 7 days of ED/NC visit - either shunt obstruction confirmed during shunt revision surgery or shunt patency confirmed by no surgery or patency confirmed in surgery - to determine Positive and Negative Predictive Value
  Interventions: Device: Imaging

INTERVENTIONS:
Device: ShuntCheck-Micro-Pumper (SCMP) — ShuntCheck uses thermal dilution to detect flow in CSF shunts. CSF is cooled transcutaneously with an ice pack and ShuntCheck's thermosensor detects a temperature drop due to CSF flow "downstream" of the ice. Micro-Pumper is a handheld device which vibrates the shunt valve to generate a temporary increase in CSF flow in patent but temporarily non-flowing shunts. This flow increase can be detected by ShuntCheck.
  Arms: SCMP Rule Out for Low Risk Cases; SCMP plus Imaging; SCMP plus Imaging in Uncertain Cases
Device: Imaging — Imaging of ventricle size
  Other Names: CT Scan; MRI
  Arms: Imaging Alone; Imaging Rule for Low Risk Cases; Imaging alone in Uncertain Cases; SCMP plus Imaging; SCMP plus Imaging in Uncertain Cases

SUMMARY:
Primary objective is to demonstrate that data collected from ShuntCheck-Micro-Pumper (SCMP) testing results can be used in conjunction with imaging to diagnose shunt patency or obstruction in pediatric/adolescent subjects presenting to an Emergency Department or Neurosurgery Clinic (ED/NC). SCMP results and SCMP results combined with other diagnostic methods, including the Attending Physician's and the Neurosurgeon's clinical judgment will be compared to clinical outcomes within 7 days of ED/NC visit - either shunt obstruction confirmed during shunt revision surgery or shunt patency confirmed by no surgery or patency confirmed in surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, older than 35 months and less than 20 years of age.
2. Parent/guardian or alert subject (age 18 or over) capable of giving consent; subject less than 18 and of assent age must give assent to participate if appropriate and required by the institution. If the subjects are incapable of giving assent, then only parent/guardian consent is required.
3. Possess an unambiguously identifiable chronically indwelling ventricular shunt which crosses the clavicle.
4. Suspicion of shunt obstruction is great enough to warrant the performance of any diagnostic test for this condition
5. Will be available for follow-up for up to 7 days

Exclusion Criteria:

1. Inability or unwillingness of the parent/guardian or alert subject to give informed consent/assent (when appropriate) as required by the Institutional Review Board.
2. Presence of multiple shunts or known non-functioning shunts crossing the clavicle.
3. Evaluating staff rule out shunt obstruction on the basis of a physical/clinical examination.
4. SCMP test would interfere with emergent subject care or if the subject is scheduled to go the OR in short order.
5. Presence of an interfering open wound or edema over the shunt.
6. Likelihood, in the judgment of the investigator, of the subject being lost to follow-up as a result of subject unavailability or clinical outcome being unobtainable.
7. Any other condition that would preclude or bias the results of the study according to the judgment of the investigator.
8. Judgment of the investigator that participation in the study will interfere with, or be detrimental to, administration of optimal health-care to the subject.

Ages: 35 Months to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-06 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy compared with clinical outcomes | 7 days
  SCMP results and SCMP results combined with other diagnostic methods, including the Attending Physician's and the Neurosurgeon's clinical judgment will be compared to clinical outcomes within 7 days of ED/NC visit - either shunt obstruction confirmed during shunt revision surgery or shunt patency confirmed by no surgery or patency confirmed in surgery.
Positive Predictive Value (PPV) | 7 days
  Specifically to demonstrate that SCMP positive (Flow Not Confirmed - FNC) plus imaging positive (enlarged ventricles) results yield a higher positive predictive value than imaging positive alone.
Negative Predictive Value (NPV) | 7 days
  Specifically to demonstrate that SCMP negative (Flow Confirmed - FC) plus imaging negative (non-enlarged ventricles) results yield a higher negative predictive value than imaging negative alone.
Safety | 1 day
  To determine if any adverse events were caused by the device or procedure while using the study device.

SECONDARY OUTCOMES:
Rule Out for Low Risk Cases | 7 days
  To demonstrate that SCMP plus Physician's judgment is comparable to Physician's judgment plus imaging in ruling out shunt malfunction in patients judged to be "Unlikely to require shunt surgery"
Increased PPV and NPV for Uncertain Cases | 7 days
  To demonstrate that SCMP plus imaging results yield higher positive and negative predictive values than imaging alone in patients who are admitted for observation.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph R Madsen, MD, Study Chair — Boston Children's Hospital; George I Jallo, MD, Principal Investigator — Johns Hopkins University; David A Frim, MD, Principal Investigator — University of Chicago Comer Children's Hospital; David Sandberg, MD, Principal Investigator — University of Texas-Houston/Children's Memorial Hermann Hospital; Phillip B Storm, MD, Principal Investigator — Children's Hospital of Philadelphia; Joseph J Zorc, MD, Principal Investigator — Children's Hospital of Philadelphia; Robert W Hickey, MD, Principal Investigator — University of Pittsburgh; Mandeep Tamber, MD, Principal Investigator — University of Pittsburgh; Lisa H Merck, MD MPH, Principal Investigator — Rhode Island Hospital; Petra M Klinge, MD PhD, Principal Investigator — Rhode Isalnd Hospital; Robert F Keating, MD, Principal Investigator — Children's National Research Institute; James Chamberlain, MD, Principal Investigator — Children's National Research Institute; Jeffrey R Leonard, MD, Principal Investigator — Nationwide Children's Hospital; Julie C Leonard, MD MPH, Principal Investigator — Nationwide Children's Hospital; Joseph H Piatt, MD, Principal Investigator — Alfred I. duPont Hospital for Children; Jonathan E Bennett, MD, Principal Investigator — Alfred I. duPont Hospital for Children; David Chesler, MD, Principal Investigator — Stony Brook Medical Center
Locations (11):
- United States (11):
  - A I dePont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Chicago Comer Children's Hospital, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Stony Brook Medical Center, Stony Brook, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Texas-Houston/Children's Memorial Hermann Hospital, Houston, Texas